CLINICAL TRIAL: NCT03174912
Title: In the Prediction of Recurrence and Progression of NMIBC; EORTC or CUETO or Both?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Muhammet Fatih Kilinc, Principal investigator, Medical doctor, Ankara Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5050
Record Dates: First submitted 2017-05-29; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Bladder Cancer; Disease Progression; Recurrent Bladder Cancer
Keywords: EORTC; CUETO; bladder neoplasm; disease progression; recurrence
MeSH Terms: conditions — Urinary Bladder Neoplasms; Disease Progression; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Whole patient group (patients not treated with BCG and patients treated with BCG)
  Interventions: Procedure: Intravesical BCG instillation
- Group 2 (No Intervention): Patients not treated with BCG
- Group 3 (Active Comparator): Patients treated with BCG
  Interventions: Procedure: Intravesical BCG instillation

INTERVENTIONS:
Procedure: Intravesical BCG instillation — ıntravesical BCG instillations were done two weeks after transurethral resection of bladder cancer
  Arms: Group 1; Group 3

SUMMARY:
Investigators aimed to evaluate the performance of The European Organization for Research and Treatment of Cancer(EORTC) and the Spanish Urology Association for Oncological Treatment(CUETO) risk tables on all non-muscle invasive bladder cancer patients(NMIBC), and those not treated with BCG and treated with BCG separately.

DETAILED DESCRIPTION:
Risk tables can be used for the prediction of recurrence and especially progression of nonmuscle invasive bladder cancer .The European Organization for Research and Treatment of Cancer(EORTC) developed a risk table,which provides a scoring system for recurrence and progression risk.The EORTC risk table includes these factors: number of tumors,tumor size,prior recurrence rate,T stage,presence of carcinoma in situ(CIS),and grade for NMIBC patients not treated by maintenance bacillus Calmette-Guerin(BCG) instillation therapy.The Spanish Urology Association for Oncological Treatment(CUETO)later proposed a modified model to be used for patients only treated with BCG instillation.This risk table includes these factors:age,gender,recurrent tumor,number of tumors,T stage,CIS,and grade.

There is no risk table that can be used for NMIBC patients treated or not treated with BCG.Should we use the EORTC risk table for patients not treated with BCG and the CUETO table only for those treated with BCG or is one of them sufficient to predict recurrence and progression in all patients?The main aim of this study was to compare the utility of the EORTC and CUETO risk tables in all patients, and separately in patients not treated with BCG and treated with BCG.

ELIGIBILITY:
Inclusion Criteria:

* primary or recurrent bladder cancer
* non-muscle invasive bladder cancer
* at least 60 months follow-up period if progression was not determined.

Exclusion Criteria:

* primary CIS,
* muscle-invasive disease after second look TUR-BT
* non-urothelial carcinoma of the bladder,
* concomitant upper urinary tract tumor,
* not able to contacted for whatever reason

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrence or progression | From date of participitant recruitment until the date of first documented progression or recurrence or death from any cause, whichever came first, assessed up to 60 months
  The primary end point for recurrence was accepted as the occurrence of the first recurrence or progression

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Xylinas E, Kent M, Kluth L, Pycha A, Comploj E, Svatek RS, Lotan Y, Trinh QD, Karakiewicz PI, Holmang S, Scherr DS, Zerbib M, Vickers AJ, Shariat SF. Accuracy of the EORTC risk tables and of the CUETO scoring model to predict outcomes in non-muscle-invasive urothelial carcinoma of the bladder. Br J Cancer. 2013 Sep 17;109(6):1460-6. doi: 10.1038/bjc.2013.372. Epub 2013 Aug 27. PMID 23982601
- [Result] Xu T, Zhu Z, Zhang X, Wang X, Zhong S, Zhang M, Shen Z. Predicting recurrence and progression in Chinese patients with nonmuscle-invasive bladder cancer using EORTC and CUETO scoring models. Urology. 2013 Aug;82(2):387-93. doi: 10.1016/j.urology.2013.04.007. Epub 2013 Jun 10. PMID 23759377